CLINICAL TRIAL: NCT04305795
Title: An Open-label Study Using ASP-1929 Photoimmunotherapy in Combination With Anti-PD1 Therapy in EGFR Expressing Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rakuten Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASP-1929-181
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Head and Neck Squamous Cell Carcinoma; Metastatic Head-and-neck Squamous-cell Carcinoma; Locally Advanced Cutaneous Squamous Cell Carcinoma; Metastatic Cutaneous Squamous Cell Carcinoma
Keywords: Rakuten Medical; ASP-1929; HNSCC; CUSCC; head and neck; cutaneous; squamous cell carcinoma; photoimmunotherapy; PIT; skin; EGFR; Anti-PD1; Pembrolizumab; Cemiplimab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — pembrolizumab; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Sub-study 1- 1L HNSCC (Other): Recurrent locally advanced and/or metastatic head and neck squamous cell carcinoma
  Interventions: Biological: 200 mg Pembrolizumab; Combination Product: ASP-1929 PIT
- Sub-study 2- 1L cuSCC (Other): Locally advanced or metastatic cutaneous squamous cell carcinoma
  Interventions: Biological: 350 mg Cemiplimab; Combination Product: ASP-1929 PIT
- Sub-study 3- 2L cuSCC (Other): Locally advanced or metastatic cutaneous squamous cell carcinoma
  Interventions: Biological: 350 mg Cemiplimab; Combination Product: ASP-1929 PIT

INTERVENTIONS:
Biological: 200 mg Pembrolizumab — every 3 weeks on Days 1 and 22 of each 6-week cycle for up to 24 months.
  Arms: Sub-study 1- 1L HNSCC
Biological: 350 mg Cemiplimab — every 3 weeks on Days 1 and 22 of each 6-week cycle for up to 24 months.
  Arms: Sub-study 2- 1L cuSCC; Sub-study 3- 2L cuSCC
Combination Product: ASP-1929 PIT — ASP-1929 IV on Day 8 of each 6-week cycle for up to 24 months.
  Photoimmunotherapy Light Treatment on Day 9 of each 6-week cycle for up to 24 months.

SUMMARY:
Open-label study using ASP-1929 photoimmunotherapy in combination with anti-PD1 therapy in patients with recurrent or metastatic head and neck and squamous cell cancer or advanced or metastatic cutaneous squamous cell carcinoma.

DETAILED DESCRIPTION:
This basket trial study has 3 sub-studies:

Sub-study 1 (181 HNSCC) will enroll patients with recurrent or metastatic (R/M) squamous cell cancer of the head and neck (HNSCC). HNSCC patients are required to have positive expression of programmed cell death ligand 1 (PD-L1) defined by Combined Positive Score (CPS) ≥1.

Sub-study 2 (181 cuSCC) will enroll patients with locally advanced or metastatic cutaneous squamous cell carcinoma (cuSCC).

Sub-study 3 (181 2LcuSCC) will enroll patients with locally advanced or metastatic cutaneous squamous cell carcinoma who have progressed on anti-PD-1 therapy.

Eligible patients will enroll in the applicable sub-study and receive ASP-1929 photoimmunotherapy (PIT) treatment in combination with an anti-PD-1 therapy for up to 24 months. During the treatment period, patients will undergo clinical assessments and be monitored for safety and tolerability and disease progression by modified RECIST 1.1 for overall response rate (ORR), progression-free survival (PFS), and duration of response (DOR).

Each sub-study is an open-label, single-arm study. For each sub-study, the primary objectives are to characterize the safety and tolerability of ASP-1929 PIT treatment in combination with anti-PD-1 treatment and to assess the effect of ASP-1929 PIT treatment with anti-PD1 therapy on tumor response.

ELIGIBILITY:
Overall Inclusion Criteria:

Provide written informed consent

• Cancers as follows:

Sub-study 1: Histologically or cytologically confirmed recurrent locally and/or metastatic head and neck squamous cell carcinoma with Combined Positive Score (CPS) ≥ 1 as determined by a CLIA certified and/or FDA approved test.

Note: A multi-disciplinary group (including a surgeon and radiation oncologist) must agree that the patient is not a candidate for locoregional therapy.

Sub-study 2: Histologically or cytologically confirmed locally advanced or metastatic cutaneous squamous cell carcinoma not amenable to definitive surgery or radiation.

Sub-study 3: Histologically or cytologically confirmed locally advanced or metastatic cutaneous squamous cell carcinoma not amendable to definitive surgery or radiation.

* At least one site of disease accessible to light illumination.
* Measurable disease by modified RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* No prior systemic therapy administered in the recurrent and/or metastatic setting (with the exception of systemic therapy completed ≥ 6 months prior if given as part of multimodal treatment for locally advanced disease). (Sub-study 1 only).
* Patients must be actively receiving single-agent, systemic anti-PD1 therapy at the time of screening (Sub-study 3 only).
* Disease progression despite at least 2 months of anti-PD1 therapy at the time of screening. Progression must be confirmed by at least two scans at least one month apart. Screening scan may serve as confirmation of progression (Sub-study 3 only).
* Adequate organ function.
* Female patients of childbearing potential must have a negative pregnancy test at screening and must be willing to use 2 methods of highly effective birth control while on study or be surgically sterile, or abstain from heterosexual sexual activity for the course of the study through 120 days after the last dose of anti-PD1 treatment.
* Male participants must agree to use a highly effective method of contraception starting with the first dose of study medication through 120 days after the last dose of anti-PD1 treatment.

Exclusion Criteria:

* Prior therapy with an anti-PD1 or anti-PD-L1 (Sub-study 1 only).
* Prior systemic therapy that is not intended as part of definitive treatment (eg, induction, concurrent, adjuvant, or neoadjuvant treatment) (Sub-studies 1 and 2 only).
* Systemic anti-PD-1 therapy prior to current course of definitive therapy (Sub-study 3 only).
* Prior systemic therapy given as definitive treatment (chemotherapy, EGFR inhibition). Patients with a history of prior chemoradiation are eligible (Sub-study 3 only).
* Radiation therapy (or other non-systemic therapy) within 4 weeks prior to study Day 1 or not fully recovered from adverse events due to a previously administered treatment
* Receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to Cycle 1 Day 1.
* Diagnosed and/or treated for additional malignancy within 2 years prior to study Day 1, except for, curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected in situ cervical and/or breast cancers.
* History of significant (≥ Grade 3) cetuximab infusion reactions.
* Prior allogeneic tissue/solid organ transplant.
* Known or active central nervous system metastases and/or carcinomatous meningitis.
* Active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
* Evidence of interstitial lung disease or current active, noninfectious pneumonitis.
* Active infection requiring systemic therapy.
* Known or active bacterial, viral, and fungal infection including tuberculosis, active Hepatitis B (eg, HBsAg reactive), or Hepatitis C (eg, RNA [qualitative] is detected)
* Known history of testing positive for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Received a live vaccine within 30 days of study Day 1. Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (eg, Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Requiring future examinations or treatments within 4 weeks after an ASP-1929 PIT treatment cycle exposing the patient to significant light (eg, eye examinations, surgical procedures, endoscopy) that is unrelated to the ASP-1929 PIT treatment
* Patients expecting to breastfeed during the study and through 120 days after the last dose of study treatment.
* Major surgery or significant traumatic injury ≤ 28 days before study day 1, or anticipation of the need for major surgery during the course of study treatment.
* Currently participating or participated in a study of an investigational agent and received study therapy (including RM-1929 or ASP-1929 PIT studies), or used an investigational device within 4 weeks of study Day 1.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Characterize the safety and tolerability of ASP-1929 PIT treatment in combination with anti-PD1 therapy | 24 months
  Treatment Emergent Adverse Events (TEAE) and Serious TEAE
HNSCC: Assess the effect of ASP-1929 PIT treatment with anti-PD1 therapy on tumor response | 24 months
  Objective Response Rate (ORR) per modified RECIST 1.1, as assessed by investigator
cuSCC: Assess the effect of ASP-1929 PIT treatment with anti-PD1 therapy on tumor response | 24 months
  Objective Response Rate (ORR) per modified RECIST 1.1, by central review of tumor imaging by photography and radiographic assessments

SECONDARY OUTCOMES:
Overall Survival (OS) | 24 months
  Assess the effect of ASP-1929 PIT treatment in combination with anti-PD1 therapy on survival
Progression-free survival (PFS) | 24 months
  Assess the effect of ASP-1929 PIT treatment in combination with anti-PD1 therapy on survival
Duration of Response (DOR) | 24 months
  Assess the effect of ASP-1929 PIT treatment in combination with anti-PD1 therapy on survival
cuSCC: Objective Response Rate (ORR) per modified RECIST 1.1, as assessed by investigator review of tumor imaging by photography and radiographic assessments | 24 months
  Assess the effect of ASP-1929 PIT treatment in combination with anti-PD1 therapy on tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki Suzuki, MD, Study Director — Rakuten Medical, Inc.
Locations (7):
- United States (7):
  - University of Miami Hospital and Clinics, Miami, Florida
  - University of Kentucky, Lexington, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Providence Medical Center, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas, MD Anderson Cancer Center, Houston, Texas